CLINICAL TRIAL: NCT03895944
Title: Phase 1, Open-label, Single-arm, Dose-escalation Clinical Study Evaluating the Safety and Efficacy of ET190L1-ARTEMIS™2 in Relapsed, Refractory B Cell Leukemia and Lymphoma
Brief Title: ET190L1-ARTEMIS™ T Cells in Relapsed, Refractory B Cell Leukemia and Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2017LSL-C001
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: CD19+ Lymphoma, B-Cell; CD19+ Leukemia, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- iv low dose (Experimental): Autologous ET190L1-ARTEMIS™ T cells administered by intravenous (IV) infusion with low dose (1x10^6) in Leukemia or Lymphoma patients
  Interventions: Biological: ET190L1-ARTEMIS™ T cells -iv low dose
- iv middle dose (Experimental): Autologous ET190L1-ARTEMIS™ T cells administered by intravenous (IV) infusion with middle dose (3x10^6) in Leukemia or Lymphoma patients
  Interventions: Biological: ET190L1-ARTEMIS™ T cells -iv middle dose
- iv high dose (Experimental): Autologous ET190L1-ARTEMIS™ T cells administered by intravenous (IV) infusion with high dose (10x10^6) in Leukemia or Lymphoma patients
  Interventions: Biological: ET190L1-ARTEMIS™ T cells - iv high dose

INTERVENTIONS:
Biological: ET190L1-ARTEMIS™ T cells -iv low dose — Autologous T cells transduced with lentivirus encoding an anti-CD19 (ET190L1) -ARTEMIS™ expression construct, 1x10^6
  Arms: iv low dose
Biological: ET190L1-ARTEMIS™ T cells -iv middle dose — Autologous T cells transduced with lentivirus encoding an anti-CD19 (ET190L1) -ARTEMIS™ expression construct, 3x10^6
  Arms: iv middle dose
Biological: ET190L1-ARTEMIS™ T cells - iv high dose — Autologous T cells transduced with lentivirus encoding an anti-CD19 (ET190L1) -ARTEMIS™ expression construct, 10x10^6
  Arms: iv high dose

SUMMARY:
Clinical study to evaluate safety and pharmacokinetics (primary objectives) and efficacy (secondary objective) of ET190L1-ARTEMIS™2 T-cells in patients with Cluster of Differentiation (CD) 19+ B cell Leukemia and Lymphoma

DETAILED DESCRIPTION:
ARTEMIS™ is a novel chimeric T-cell therapy that in pre-clinical studies, functionally matches the efficacy of Chimeric Antigen Receptor (CAR) T cells, but dramatically reduces the release of cytokines upon killing of target positive tumors. The molecular target for ET190L1-ARTEMIS™ is Cluster of Differentiation 19 (CD19), which is expressed on B cell Lymphomas and B cell Leukemias. ET190L1-ARTEMIS™ is a second generation ARTEMIS™ receptor engineered with a human Fab antibody domain against CD19. This clinical study evaluates the safety and pharmacokinetics of ET190L1-ARTEMIS™ T-cells in patients with relapsed/refractory B-cell lymphoma and B-cell Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory CD19+ B-cell lymphoma or Leukemia, with no effective therapy available per National Comprehensive Cancer Network (NCCN) guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2, expected survival time > 3 months per PIs opinion
* Women of childbearing age should have a negative pregnancy test and agree to use effective contraception during treatment and 1 year after the last dose.
* Peripheral venous access is available and no issues with apheresis for lymphocyte isolation
* serum alanine aminotransferase(ALT)<200 Unit/L, ALT/Aspartate aminotransferase(AST)<3 normal range; serum creatinine (Cr)<2.5mg/dL
* Voluntarily signed informed consent form

Exclusion Criteria:

* Women in pregnancy and lactation
* Unable to perform leukapheresis and iv infusion
* With active infection
* Major organ failure
* Patients with dependence on corticosteroids
* Continuously used glucocorticoids or other immunosuppressive agents within 2 weeks
* T cell deficiency or T cells are difficult to be transduced
* Patients currently receiving other investigational treatments (biotherapy, chemotherapy, or radiotherapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-12-06 (Estimated); Study Completion 2019-12-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of ARTEMIS T cell treatment-related adverse events | until 24 weeks
  Frequency of treatment-related adverse events that occurred at any time from the first day of infusion that are "possibly", "likely", or "definitely" related to the study, including infusion related toxicity and ET190L1-ARTEMIS™ T T cells related toxicity. Include but not limited to: Fever, chills, nausea, vomiting, jaundice and other gastrointestinal symptoms; Fatigue, hypotension, respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction. Assessed at all visits.
Number of ET190L1-ARTEMIS™ T cells in peripheral blood | 24 months
  Duration of in vivo engraftment of ET190L1-ARTEMIS™ T cells. Number of ET190L1-ARTEMIS™ T cells in peripheral blood will be presented as Time to peak, Time to baseline level and so on.
% of ET190L1-ARTEMIS™ T cells in peripheral blood | 24 months
  Duration of in vivo engraftment of ET190L1-ARTEMIS™ T cells. % of ET190L1-ARTEMIS™ T cells in peripheral blood will be presented as Time to peak, Time to baseline level and so on.
Maximum Tolerated Dose | 28 days up to 2 years
  Determine the safety, including potential dose limiting toxicities, of the ET190L1-ARTEMIS™ T cells. A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the ET190L1-ARTEMIS™ T cells, which is irreversible or life threatening or CTCAE Grade 3-5. Assessed at all visits.

SECONDARY OUTCOMES:
Tmax of serum cytokine levels | 24 weeks
  Increase or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immunoassays will be presented as time to peak level.
Time to baseline for serum cytokine levels | 24 weeks
  Increase or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immunoassays will be presented as time to baseline.
AUC of serum cytokine levels | 24 weeks
  Increase or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immunoassays will be presented as area under curve (AUC).
Rate of disease response | 28 days to 24 months
  Rate of disease response assessed by Lugano classification (a lymphoma staging classification). Response rates will be estimated as the percent of patients with any of the following: complete remission (CR), partial response (PR).
Progression free survival (PFS) | 4 months, 1 year and 2 years
  Progression free survival (PFS)
Median Survival（MS） | 4 months, 1 year and 2 years
  Median Survival（MS）
Overall Survival（OS） | 4 months, 1 year and 2 years
  Overall Survival（OS）
B cell depletion (Number) | 2 years
  Number of B cells in peripheral blood will be presented as time to baseline level and time to recover for up to 2 years.
B cell depletion (%) | 2 years
  % of B cells in peripheral blood will be presented as time to baseline level and time to recover for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Zhang, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China